CLINICAL TRIAL: NCT06797713
Title: The Effect of Perioperative Targeted Fluid Therapy on Postoperative Cognitive Dysfunction in Coronary Artery Bypass Surgery.
Brief Title: Effect of Targeted Fluid Therapy on Postoperative Cognitive Dysfunction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gamze Talih, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/282
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Dysfunction, Postoperative
Keywords: Goal-directed fluid treapy; Postoperative cognitive dysfunction; Coronary artery bypass graft surgery; conventional fluid therapy
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Intervention Model Description: All patients will have a Montreal cognitive assessment questionnaire (MOKA) for cognitive dysfunction one day before the operation and blood will be taken to the biochemistry tube to study NLRP3, IL-18, IL-1 beta and caspase 1 simultaneously. In the group where targeted fluid therapy will be applied (Group D,n=30), esophageal doppler will be placed, fluid, inotropes, blood replacements will be made according to the recommendations of the guidelines on this subject (such as stroke volume, SVV, oxygen delivery, etc.). Patients in the control group (Group C, n=30) will receive fluid and blood product treatment by following standard parameters (blood pressure, urine output, serum lactate level, base excess). Delirium will be monitored with the confusion assessment method every day for 7 days postoperatively. The MOKA test will be repeated on the 7th and 30th days postoperatively,blood samples will be taken and NLRP-3, IL-1 beta, IL-18, caspase-1 will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (D): Doppler Group (Active Comparator): Patient group receiving targeted fluid therapy with esophageal doppler
  Interventions: Procedure: Esophageal doppler
- Group (C): Control Group (Sham Comparator): Group of patients receiving conventional fluid therapy
  Interventions: Procedure: Conventional method

INTERVENTIONS:
Procedure: Esophageal doppler — Fluid/inotrope decisions will be made with parameters such as stroke volume (SV), stroke volume variation (SVV), pulse pressure variation (PVV), systemic vascular resistance (SVR), and cardiac output (CO) on the Doppler monitor screen.
  Arms: Group (D): Doppler Group
Procedure: Conventional method — Fluid therapy is performed by monitoring parameters such as blood pressure, urine output, lactate...
  Arms: Group (C): Control Group

SUMMARY:
Postoperative cognitive dysfunction (POCD) describes a decline in cognitive function as measured by pre- and postoperative neuropsychological testing. It is common after cardiac surgery, affecting 25% to 70% of patients, and is usually associated with pathophysiological mechanisms such as cerebral hypoperfusion, cerebral microemboli, glycaemic control and neurotoxic effects of anaesthetic agents. There are similar mechanisms between POCD and postoperative delirium (POD), both of which promote neuroinflammation through systemic inflammation and blood-brain barrier dysfunction. It has also been associated with concentrations of peripheral inflammatory markers (such as CRP, IL-6). The aim of this study was to examine the pathophysiological processes leading to cognitive dysfunction after cardiac surgery and to evaluate the role of targeted fluid therapy in these conditions. Targeted fluid therapy aims to optimise fluid, inotrope and vasopressor therapy by monitoring haemodynamic parameters (stroke volume, cardiac output, systemic vascular resistance, etc.).

This treatment may improve tissue perfusion, reduce the inflammatory response and reduce mortality. In this study, the optimisation of fluid therapy during cardiac surgery was achieved by using monitors based on oesophageal doppler and pulse contour analysis. The effectiveness of these methods in reducing major complications and improving clinical outcomes will be evaluated.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is cognitive dysfunction defined as a decline in cognitive function from baseline performance as measured by neuropsychological tests before and after surgery. Perioperative neurocognitive impairment includes preoperative neurocognitive impairment, POCD and postoperative delirium (POD). It is extremely common after cardiac surgery and affects 25% to 70% of patients. The underlying pathophysiological mechanisms leading to cognitive impairment are unclear, but many factors have been implicated in the aetiology. Pathophysiological mechanisms leading to cognitive dysfunction following cardiac surgery such as cerebral hypoperfusion, cerebral microemboli, glycaemic control and possible neurotoxic effects of anaesthetic agents have been demonstrated in the literature. The increase in the frequency of neurocognitive impairments leads to prolonged hospitalisation and increased healthcare costs. Although there are many clinical differences between POD and POCD, both lead to blood-brain barrier dysfunction and promote neuroinflammation through a systemic inflammatory response triggered by surgical trauma.

It has been shown that NOD-LRR- and pyrin domain-containing protein 3 (NLRP3) increased in the hippocampus of mice after cardiac surgery, causing hippocampal inflammation and cognitive dysfunction. In another study, it was reported that microglia in the hippocampus of rats were activated, the amount of inflammatory factors such as IL-1β, IL-6 and TNF-α increased and the permeability of the blood-brain barrier increased. POD and POCD were also found to be closely related with the concentration of peripheral inflammatory markers (such as CRP, IL-6).

Targeted fluid therapy (TFT) in cardiac surgery is the use of various haemodynamic parameters (e.g. stroke volume, cardiac output, systemic vascular resistance and stroke volume variation) and optimisation of fluids, inotropes and vasopressors to ensure adequate tissue perfusion. Because administration of more or less fluid and blood products than needed will cause many undesirable clinical conditions in patients (in case of over administration; pulmonary oedema, tissue oedema, connective and mucosal oedema or in case of under administration; perfusion failure in peripheral tissue and brain, hypotension). The aim of targeted fluid therapy is to use haemodynamic parameters that allow us to monitor the amount of fluid, inotrope requirement, tissue blood flow and oxygenation. This optimization reduces mortality by providing normal tissue perfusion, preventing inflammatory response and possible fatal complications. There are many monitors on the market that have developed rapidly in recent years and are now used in many anaesthesia clinics for perioperative volume management. When choosing this, the aim should be to select the technology that provides the most accurate and relevant haemodynamic data, taking into account the safety, comfort and general care of the patient.

For targeted fluid therapy, techniques/monitors routinely used in clinics that have them include PiCCO plus, FloTrac/EV1000, oesophageal doppler and pulmonary artery catheter. In a study conducted in major abdominal surgeries, patients followed up with Vigileo/FloTrac, which uses the principle of oesophageal doppler and pulse contour analysis for targeted fluid therapy, were compared and it was shown that major complications and mortality decreased and it was reported that the monitors were cost effective . The fact that the sternum is open in cardiac surgery is an important limitation of monitors working on the principle of pulse contour analysis. Therefore, in this study, we planned to perform advanced haemodynamic monitoring with oesophageal Doppler and to decide on fluid/blood/inotrope support by using many parameters such as stroke volume, cardiac index, oxygen delivery, and stroke volume variation (SVV) on this monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo coronary artery bypass surgery.

Exclusion Criteria:

* Exclusion criteria are the same for both groups.

  1. Patients with mental disorders or neurological diseases.
  2. Illiterate people
  3. Patients who use medication that affects cognitive function
  4. Emergency surgeries
  5. Patients with end-stage renal failure
  6. Patients who are receiving antidepressant and antipsychotic treatment
  7. Patients who refused to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive disfunction | The evaluation will be completed 4 weeks after the intraoperative TFT.
  TFT affects postoperative cognitive dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Melikgazi, Kayseri, Turkey (Türkiye)